CLINICAL TRIAL: NCT00389844
Title: Testing the Effectiveness of the Exercise Plus Program on Efficacy Expectations, Exercise Behavior & Activity of Older Adults Following a Hip Fracture
Brief Title: BHS5 - Testing the Effectiveness of the Exercise Plus Program
Acronym: Hip5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jay S. Magaziner, Chair, Department Of Epidemiology & Public Health; Director, Center For Research On Aging, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H-22361; 5R01AG017082-04 (NIH)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Hip Fracture
Keywords: hip fracture; exercise; motivation
MeSH Terms: conditions — Hip Fractures; Motor Activity | interventions — Exercise; Elements; Information Motivation Behavioral Skills Model

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): Routine care
- 2 (Active Comparator): Exercise only
  Interventions: Behavioral: Exercise Trainer component of the Exercise Plus Program
- 3 (Active Comparator): Motivation only
  Interventions: Behavioral: Exercise Trainer component of the Exercise Plus Program; Behavioral: Plus component (motivation) of the Exercise Plus Program
- 4 (Experimental): Exercise plus motivation
  Interventions: Behavioral: Exercise Trainer component of the Exercise Plus Program; Behavioral: Plus component (motivation) of the Exercise Plus Program; Behavioral: Exercise Plus Program (exercise + motivation)

INTERVENTIONS:
Behavioral: Exercise Trainer component of the Exercise Plus Program — With the exception of the routine care group, the exercise trainers visited each of the participant in their homes twice a week for two months, once a week for four months, and once a month for six months.
  Other Names: Exercise
  Arms: 2; 3; 4
Behavioral: Plus component (motivation) of the Exercise Plus Program — Motivation only
  Other Names: Motivation
  Arms: 3; 4
Behavioral: Exercise Plus Program (exercise + motivation) — Exercise plus motivation
  Other Names: Exercise; Motivation
  Arms: 4

SUMMARY:
The major goals of this study are:

To implement a self-efficacy based intervention to strengthen efficacy beliefs related to exercise, decrease perceived barriers to exercise, and increase exercise behavior and overall activity of older women who have sustained a hip fracture.

To test the effectiveness of the Exercise Trainer component of the intervention on exercise behavior, activity, efficacy expectations, barriers to exercise, performance behaviors, overall health status, mood, pain, fear of falling, falls and fall-related injuries at 2, 6, and 12 months following fracture.

DETAILED DESCRIPTION:
Hip fracture is a major public health problem with striking consequences for the older adult, his or her family, and the health care system. By the year 2040, over 650,00 hip fractures will occur annually in older adults over the age 65. Many surviving the hip fracture will have decreased functional performance and be unable to live independently in the community. Moreover, the greatest loss in bone density and muscle strength occurs in the first two months post hip fracture. Recovery following a hip fracture has been shown to be greatly facilitated by participation in a rehabilitation program, and continued participation in a regular exercise program can increase functional recovery, muscle strength, and prevent future fractures. Despite the benefits of exercise, it is difficult to initiate exercise activity in older adults, and helping them adhere to an exercise regime is even more challenging. Self-efficacy, a belief in the individual's capabilities to perform a course of action to attain a desired outcome, and outcome expectancy, the belief that carrying out behavior will lead to a desired outcome, are hypothesized to be critical factors in adhering to a regular exercise program.

A total of 240 subjects (60 per group) from five area hospitals meeting the eligibility criteria will be recruited into the study. A study nurse will periodically contact a designated liaison at each hospital to obtain the names of patients with hip fractures. Following identification, a study nurse will contact the patient to enroll them in the study.

An experimental 2 X 2 factorial design with repeated measures will be used to test the impact of a self-efficacy based intervention on exercise behavior, activity, efficacy beliefs and barriers, performance, health status, mood, falls, fear of falling, and fall-related injuries of older adults who sustained a hip fracture.

Participants will be randomized after consent is obtained and the baseline evaluation completed. Participants will be randomly assigned to one of the four groups defined by the 2 X 2 design: (1) the Exercise Only component (2) the Plus (motivation) component; (3) Exercise Plus (exercise + motivation) components, and (4) routine care.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture

Exclusion Criteria:

* Male
* Under 65 years old
* Non-community dwelling
* Fractured more than 72 hours before admission to the hospital
* Pathologic fracture
* Resides more than 70 from the hospital of admission
* Recent diagnosis (in past 6 months) of angina or myocardial infarction
* Myocardial infarction or stroke concurrent with hip fracture
* Diagnosis of ventricular arrhythmia, third degree heart block, atrial fibrillation or if vital signs=heart <60 or >100
* Active or suspected myocarditis or pericarditis in the past year
* Recent (within past 6 months) deep venous thrombosis or intracardiac thrombi
* Persistent pulmonary edema during hospitalization
* Poorly controlled blood pressure w/ resting systolic >180 mm Hg or resting diastolic >100 mm Hg (3 or more readings with 24-hour period)
* Presence of ventricular aneurysm
* Paget's Disease
* Diabetes with blood sugar consistently > 300
* Diagnosis of thyrotoxicosis or myxedema within past year
* Any diagnosis of hyperparathyroidism, hypoparathyroidism, or osteomalacia
* Parkinson's, multiple sclerosis, or ALS (Lou Gehrig's disease)
* New (past 6 months) onset seizure disorder or seizure within the past 6 months
* Diagnosis of schizophrenia
* Recent (within past 6 months) GI hemorrhage or bleeding
* Preadmission coumadin therapy
* Cirrhosis or end stage renal disease (ESRD)
* Advanced hepatitis, AIDS, or endocarditis
* Cancer with metastases, or cancer under active treatment (chemotherapy with cytotoxic agents) other than non-melanomic skin cancers
* Current diagnosis of chronic alcohol abuse
* Preadmission narcotic use or preadmission benzodiazepine use more than 1 dose or tablet a day
* Required human assistance to walk prior to fracture
* Chest pains when climbing a flight of stairs, while walking on level ground, or at rest prior to the hip fracture
* Use of supplemental oxygen prior to fracture
* Other (Non-English speaking, severe blindness, paraplegia, hemiplegia
* Mini-Mental Status Exam score <20

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Actual)
Dates: Start 2000-07; Primary Completion 2004-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | 2, 6, and 12 months post hip fracture
Exercise behavior and activity | 2, 6, and 12 months post hip fracture
Subjective report of exercise | 2, 6, and 12 months post hip fracture

SECONDARY OUTCOMES:
Falls | 2, 6, and 12 months post hip fracture
Fall-related injuries | 2, 6, and 12 months post hip fracture
Fear of falling | 2, 6, and 12 months post hip fracture
Pain | 2, 6, and 12 months post hip fracture
36-item short-form health survey (SF-36) | 2, 6, and 12 months post hip fracture
Depression | 2, 6, and 12 months post hip fracture

CONTACTS AND LOCATIONS:
Overall Officials: Jay Magaziner, Ph.D., MSHyg, Principal Investigator — University of Maryland, Baltimore
Locations (5):
- United States (5):
  - Greater Baltimore Medical Center (GBMC), Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - St. Agnes Hospital, Baltimore, Maryland
  - Franklin Square Hospital, Baltimore, Maryland
  - North Arundel Hospital, Glen Burnie, Maryland

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134